CLINICAL TRIAL: NCT03301415
Title: A Phase II, Single Stage, Single-Arm Investigation of Oral Valganciclovir Therapy in Infants With Asymptomatic Congenital Cytomegalovirus Infection
Brief Title: Asymptomatic Congenital CMV Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety signal
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-0095
Record Dates: First submitted 2017-09-28; First posted 2017-10-04 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2018-10

CONDITIONS: Congenital Cytomegalovirus Infection
Keywords: Asymptomatic; Congenital CMV Infection; Valganciclovir Therapy
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Confirmed congenital CMV without baseline SNHL (Experimental): Valganciclovir 16 mg/kg/dose orally twice daily for four months, n=229
  Interventions: Drug: Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir — Valganciclovir, 16 mg/kg/dose given orally twice daily for four months

SUMMARY:
This is a phase II, open-label trial to evaluate valganciclovir as a treatment to prevent development of sensorineural hearing loss (SNHL) in infants with asymptomatic congenital cytomegalovirus (CMV) infection. The trial will be conducted in two phases - screening of newborns to identify eligible subjects, and treatment of those newborns who have confirmed CMV infection at birth but without outward manifestations of congenital CMV infection. 229 newborns with confirmed CMV infection but without baseline SNHL and who meet all inclusion/exclusion criteria will be enrolled into the treatment phase. Study duration is 5 years. Primary objective of this study is to estimate the proportion of subjects with asymptomatic congenital CMV infection who, following treatment with 4 months of oral valganciclovir, develop SNHL by 6 months of life.

DETAILED DESCRIPTION:
This is a phase II, open-label trial to evaluate valganciclovir as a treatment to prevent development of sensorineural hearing loss (SNHL) in infants with asymptomatic congenital cytomegalovirus (CMV) infection. The trial will be conducted in two phases - screening of newborns to identify eligible subjects, and treatment of those newborns who have confirmed CMV infection at birth but without outward manifestations of congenital CMV infection. Approximately 48,250 newborn infants with no outward manifestations of congenital CMV infection will be screened to detect approximately 241 neonates with asymptomatic congenital CMV infection; these 241 newborns then will have audiology examinations to determine baseline hearing, with approximately 229 having normal hearing in both ears. Those 229 newborns with confirmed CMV infection but without baseline SNHL and who meet all inclusion/exclusion criteria will be enrolled into the treatment phase. Enrolled subjects will be treated for four months with oral valganciclovir (16 mg/kg/dose, administered two times per day). Audiologic assessments will be made during the Screening Period and Study Months 4 (end of treatment), 6, 12, and 18. Treated infants will be followed for safety throughout the first 6 months of the study (including for 2 months post-treatment). Study duration is 5 years. Primary objective of this study is to estimate the proportion of subjects with asymptomatic congenital CMV infection who, following treatment with 4 months of oral valganciclovir, develop sensorineural hearing loss (SNHL) by 6 months of life. Secondary objectives are to: 1) define the safety and tolerability of valganciclovir in enrolled subjects, 2) estimate the proportion of subjects with asymptomatic congenital CMV infection who, following treatment with 4 months of oral valganciclovir, develop SNHL over the first 18 months of life.

ELIGIBILITY:
Inclusion Criteria:

* Parent(s)/legal guardian(s) have signed informed consent documents*
* Confirmation of cytomegalovirus (CMV) by urine polymerase chain reaction (PCR) testing
* Infant </= 30 days of age at initiation of study drug
* Weight at study enrollment >/= 1775 grams
* Gestational age >/= 32 weeks at birth

  * There is a screening informed consent for screening phase of study participation, and a treatment informed consent for treatment phase of study participation.

Exclusion Criteria:

* Symptomatic congenital cytomegalovirus (CMV) disease*
* Sensorineural hearing deficits as detected by formal brainstem evoked response (not a screening auditory brainstem response (abr)) of known etiology other than CMV
* Prior or current receipt of ganciclovir, valganciclovir, foscarnet, cidofovir, brincidofovir, maribavir, or letermovir
* Maternal receipt of CMV hyperimmune globulin during pregnancy
* Breastfeeding from mother who is receiving ganciclovir, valganciclovir, foscarnet, cidofovir, brincidofovir, maribavir, or letermovir
* Gastrointestinal abnormality which might preclude absorption of an oral medication (e.g., a history of necrotizing enterocolitis)
* Infants known to be born to women who are HIV positive (HIV testing is not required for study entry)
* Current receipt of other investigational drugs

  * Symptomatic disease is defined as one or more of the following: 1) thrombocytopenia, if known; 2) petechiae; 3) hepatomegaly; 4) splenomegaly; 5) intrauterine growth restriction; 6) hepatitis (elevated transaminases and/or direct bilirubin), if known; 7) central nervous system involvement of the CMV disease (such as microcephaly; radiographic abnormalities indicative of CMV CNS disease, if known; abnormal CSF indices for age, if known; chorioretinitis, if known; and/or positive CMV PCR from CSF, if known).

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Alabama - Children's of Alabama - Clinical Virology, Birmingham, Alabama
  - Arkansas Children's Hospital - Infectious Diseases, Little Rock, Arkansas
  - University of Louisville School of Medicine - Norton Children's Hospital - Infectious Diseases, Louisville, Kentucky
  - University of Mississippi - Children's Infectious Diseases, Jackson, Mississippi
  - Washington University School of Medicine in St. Louis - Center for Clinical Studies, St Louis, Missouri
  - Carolinas Medical Center - Pediatrics - Infectious Diseases, Charlotte, North Carolina
  - Nationwide Children's Hospital - Neonatology - Center for Perinatal Research, Columbus, Ohio
  - Children's Hospital of Pittsburgh of UPMC - Pediatric Infectious Diseases, Pittsburgh, Pennsylvania
  - Texas Medical Center - Texas Children's Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female infants with asymptomatic congenital CMV infection were recruited at participating sites between 20Aug2019 and 09SEP2020.
Groups:
- Confirmed Congenital CMV Without Baseline SNHL: Valganciclovir, 16 mg/kg/dose given orally twice daily for four months
Period: Overall Study
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Started | 7
Completed | 3
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Unable to comply with visit schedule | 2

BASELINE CHARACTERISTICS:
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 25.7 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Developing Sensorineural Hearing Loss (SNHL) in at Least One Ear Between Baseline and Study Month 6
Description: Audiologic assessments were made during the Screening Period and Study Months 4 (end of treatment), 6, 12, and 18. A single, independent study audiologist assessed the audiology test battery for each subject and assigned each ear the classifications of normal hearing, mild hearing loss, moderate hearing loss, severe hearing loss, or profound hearing loss based upon their hearing thresholds (in decibels). SNHL between baseline and Study Month 6 is defined as both ears with normal hearing at baseline, then at least one ear with sensorineural hearing loss (SNHL) at the 6 month follow-up.
Time Frame: Between baseline and study month 6
Population: All participants who have received at least one dose of study product and with a normal baseline hearing assessment for both ears and with hearing assessment result available at Study month 6 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 2
Participants | 0

2. Secondary Outcome: Number of Participants With Absolute Neutrophil Counts Below 500/mm^3
Description: Blood was collected for assessments of hematology and absolute neutrophil count was assessed at each study visit through Month 5
Time Frame: Day 1 through Study month 5
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 7
Participants | 1

3. Secondary Outcome: Number of Participants With Adverse Events Leading to Permanent Discontinuation of Valganciclovir Therapy, or Any Adverse Event That is Not Recovered / Not Resolved
Description: A count of participants discontinued from valganciclovir therapy due to adverse events were reported during the therapy period, and the count of participants with adverse events not recovered/not resolved were reported throughout the adverse event period.
Time Frame: Day 1 through Study month 6
Population: All participants who have received at least one dose of study product and for whom any data on safety are available.
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 7
Participants
  AEs leading to discontinuation | 1
  AEs not recovered/resolved | 4

4. Secondary Outcome: Number of Participants With Grade 3 or Higher Safety Laboratory Adverse Events
Description: At each study visit from the receipt of first dose of study drug and continuing through four weeks following the final dose of study drug, the participants were assessed for any adverse events. Lab parameters included ALT, creatinine, direct bilirubin, white blood cell count with differential, hemoglobin, platelets count. Abnormal laboratory values were reported as an AE if they worsened in severity from baseline, per the grading definitions provided in the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events.
Time Frame: From day 1 through study month 6
Population: All participants who have received at least one dose of study product and for whom any safety data are available.
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 7
Participants | 4

5. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Serious adverse events were those defined as: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, a congenital anomaly/birth defect, or were important medical events that may not result in death, be life-threatening, or require hospitalizations may be considered serious when, based upon appropriate medical judgment they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: From day 1 through study month 6
Population: All participants who have received at least one dose of study product and for whom any safety data are available.
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 7
Participants | 0

6. Secondary Outcome: Number of Participants With Grade 3 or Higher Unsolicited Adverse Events Assessed by Adapted From DAIDS Toxicity Tables
Description: as for outcome 4
Time Frame: From day 1 through study month 6
Population: All participants who have received at least one dose of study product and for whom any safety data are available.
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 7
Participants | 4

7. Secondary Outcome: Number of Participants With Mild Worsened Hearing, Represented by the Ear That Has the Larger Degree of Worsening
Description: Audiologic assessments were made during the Screening Period and Study Months 4 (end of treatment), 6, 12, and 18. A single, independent study audiologist assessed the audiology test battery for each participant and assigned each ear the classifications of normal hearing, mild hearing loss, moderate hearing loss, severe hearing loss, or profound hearing loss based upon their hearing thresholds (in decibels). SNHL between baseline and Study Month 18 is defined as both ears with normal hearing at baseline, then at least one ear with sensorineural hearing loss (SNHL) at the 18 month follow-up.
Time Frame: Screening and Study Months 4, 6, 8 and 12
Population: All participants who have received at least one dose of study product and with a normal baseline hearing assessment for both ears and with hearing assessment result available at Study month 12 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 7
Participants
  Screening | 0
  Month 4: number analyzed (Participants) | 5
  Month 4 | 0
  Month 6: number analyzed (Participants) | 2
  Month 6 | 0
  Month 8: number analyzed (Participants) | 2
  Month 8 | 0
  Month 12: number analyzed (Participants) | 1
  Month 12 | 0

8. Secondary Outcome: Number of Participants With Moderate Worsened Hearing, Represented by the Ear That Has the Larger Degree of Worsening
Description: Audiologic assessments were made during the Screening Period and Study Months 4 (end of treatment), 6, 12, and 18. A single, independent study audiologist assessed the audiology test battery for each subject and assigned each ear the classifications of normal hearing, mild hearing loss, moderate hearing loss, severe hearing loss, or profound hearing loss based upon their hearing thresholds (in decibels). SNHL between baseline and Study Month 18 is defined as both ears with normal hearing at baseline, then at least one ear with sensorineural hearing loss (SNHL) at the 18 month follow-up.
Time Frame: Screening and Study Months 4, 6, 8 and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 7
Participants
  Screening | 0
  Month 4: number analyzed (Participants) | 5
  Month 4 | 0
  Month 6: number analyzed (Participants) | 2
  Month 6 | 0
  Month 8: number analyzed (Participants) | 2
  Month 8 | 0
  Month 12: number analyzed (Participants) | 1
  Month 12 | 0

9. Secondary Outcome: Number of Participants With Profound Worsened Hearing, Represented by the Ear That Has the Larger Degree of Worsening
Description: as for outcome 7
Time Frame: Study Months 4, 6, 8 and 12
Population: All participants who have received at least one dose of study product and with a normal baseline hearing assessment for both ears and with hearing assessment result available at Study month 18 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 7
Participants
  Screening | 0
  Month 4: number analyzed (Participants) | 5
  Month 4 | 0
  Month 6: number analyzed (Participants) | 2
  Month 6 | 0
  Month 8: number analyzed (Participants) | 2
  Month 8 | 0
  Month 12: number analyzed (Participants) | 1
  Month 12 | 0

10. Secondary Outcome: Number of Participants With Severe Worsened Hearing, Represented by the Ear That Has the Larger Degree of Worsening
Description: as for outcome 7
Time Frame: Study Months 4, 6, 8 and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 7
Participants
  Screening | 0
  Month 4: number analyzed (Participants) | 5
  Month 4 | 0
  Month 6: number analyzed (Participants) | 2
  Month 6 | 0
  Month 8: number analyzed (Participants) | 2
  Month 8 | 0
  Month 12: number analyzed (Participants) | 1
  Month 12 | 0

11. Secondary Outcome: Number of Participants With Sensorineural Hearing Loss in at Least One Ear Through Study Month 4
Description: Audiologic assessments were made during the Screening Period and Study Months 4 (end of treatment), 6, 12, and 18. A single, independent study audiologist assessed the audiology test battery for each participant and assigned each ear the classifications of normal hearing, mild hearing loss, moderate hearing loss, severe hearing loss, or profound hearing loss based upon their hearing thresholds (in decibels). SNHL between baseline and Study Month 4 is defined as both ears with normal hearing at baseline, then at least one ear with sensorineural hearing loss (SNHL) at the 4 month follow-up.
Time Frame: Between screening and study month 4
Population: All participants who have received at least one dose of study product and with a normal baseline hearing assessment for both ears and with hearing assessment result available at Study month 4 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 5
Participants | 0

12. Secondary Outcome: Number of Participants With Sensorineural Hearing Loss in at Least One Ear Through Study Month 12
Description: Audiologic assessments were made during the Screening Period and Study Months 4 (end of treatment), 6, 12, and 18. A single, independent study audiologist assessed the audiology test battery for each participant and assigned each ear the classifications of normal hearing, mild hearing loss, moderate hearing loss, severe hearing loss, or profound hearing loss based upon their hearing thresholds (in decibels). SNHL between baseline and Study Month 12 is defined as both ears with normal hearing at baseline, then at least one ear with sensorineural hearing loss (SNHL) at the 12 month follow-up.
Time Frame: Between screening and study month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 1
Participants | 0

13. Secondary Outcome: Number of Participants With Sensorineural Hearing Loss in at Least One Ear Through Study Month 18
Description: as for outcome 7
Time Frame: Between screening and study month 18
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 1
Participants | 0

14. Secondary Outcome: Number of Participants With Transaminase Elevation During Treatment > / = 2 Times the Baseline Value
Description: Blood was collected for assessments of clinical chemistry and alanine aminotransferase (ALT) was assessed at screening, week 2, Week 4, Week 6, Week 8, Week 10, Week 12, Month 4, Month 5, and Month 6
Time Frame: Baseline, weeks 2, 4, 6, 8, 10, 12, months 4, 5 and 6.
Population: All participants who have received at least one dose of study product and for whom with any alanine aminotransferase result available from Day 1 through Month 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 7
Participants | 0

15. Secondary Outcome: Number of Ears of Mild Worsened Hearing
Description: Audiologic assessments were made during the Screening Period and Study Months 4 (end of treatment), 6, 12, and 18. A single, independent study audiologist assessed the audiology test battery for each participant and assigned each ear the classifications of normal hearing, mild hearing loss, moderate hearing loss, severe hearing loss, or profound hearing loss based upon their hearing thresholds (in decibels).
Time Frame: Screening and Study Months 4, 6, 12, and 18
Population: All participants who have received at least one dose of study product and with a normal baseline hearing assessment for both ears and with hearing assessment result available at Study months 4, 6, 12, 18.
Measure: Number; unit: Ears
Units Other Than Participants: Ears
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 5
Number analyzed (Ears) | 10
Ears
  Month 4 | 0
  Month 6: number analyzed (Participants) | 2
  Month 6: number analyzed (Ears) | 4
  Month 6 | 0
  Month 12: number analyzed (Participants) | 2
  Month 12: number analyzed (Ears) | 4
  Month 12 | 0
  Month 18: number analyzed (Participants) | 1
  Month 18: number analyzed (Ears) | 2
  Month 18 | 0

16. Secondary Outcome: Number of Ears of Moderate Worsened Hearing
Description: as for outcome 15
Time Frame: Screening and Study Months 4, 6, 12, and 18
Population: as for outcome 15
Measure: Number; unit: Ears
Units Other Than Participants: Ears
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 5
Number analyzed (Ears) | 10
Ears
  Month 4 | 0
  Month 6: number analyzed (Participants) | 2
  Month 6: number analyzed (Ears) | 4
  Month 6 | 0
  Month 12: number analyzed (Participants) | 2
  Month 12: number analyzed (Ears) | 4
  Month 12 | 0
  Month 18: number analyzed (Participants) | 1
  Month 18: number analyzed (Ears) | 2
  Month 18 | 0

17. Secondary Outcome: Number of Ears of Profound Worsened Hearing
Description: as for outcome 15
Time Frame: Screening and Study Months 4, 6, 12, and 18
Population: as for outcome 15
Measure: Number; unit: Ears
Units Other Than Participants: Ears
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 5
Number analyzed (Ears) | 10
Ears
  Month 4 | 0
  Month 6: number analyzed (Participants) | 2
  Month 6: number analyzed (Ears) | 4
  Month 6 | 0
  Month 12: number analyzed (Participants) | 2
  Month 12: number analyzed (Ears) | 4
  Month 12 | 0
  Month 18: number analyzed (Participants) | 1
  Month 18: number analyzed (Ears) | 2
  Month 18 | 0

18. Secondary Outcome: Number of Ears of Severe Worsened Hearing
Description: as for outcome 15
Time Frame: Screening and Study Months 4, 6, 12, and 18
Population: as for outcome 15
Measure: Number; unit: Ears
Units Other Than Participants: Ears
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
Number analyzed (Participants) | 5
Number analyzed (Ears) | 10
Ears
  Month 4 | 0
  Month 6: number analyzed (Participants) | 2
  Month 6: number analyzed (Ears) | 4
  Month 6 | 0
  Month 12: number analyzed (Participants) | 2
  Month 12: number analyzed (Ears) | 4
  Month 12 | 0
  Month 18: number analyzed (Participants) | 1
  Month 18: number analyzed (Ears) | 2
  Month 18 | 0

ADVERSE EVENTS:
Time Frame: All AEs occurring from Study Day 1 through four weeks following the last four weeks following the last dose of study drug and laboratory AEs occurring through Study Month 6 were collected.
Arm/Group | Confirmed Congenital CMV Without Baseline SNHL
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Confirmed Congenital CMV Without Baseline SNHL (N=7)
Anaemia (Blood and lymphatic system disorders) | 3 (7)
Neutropenia (Blood and lymphatic system disorders) | 7 (10)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Bilirubin conjugated increased (Investigations) | 5 (5)
Haemoglobin decreased (Investigations) | 1 (1)
Monocyte count increased (Investigations) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was stopped early due to low accrual with only 7 participants enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT03301415/Prot_SAP_002.pdf
  • Informed Consent Form (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT03301415/ICF_003.pdf